CLINICAL TRIAL: NCT04046874
Title: Implementation of a Stratified Model of Care for Low Back Pain Patients in Primary Care Settings
Brief Title: Stratified Primary Care for Low Back Pain
Acronym: SPLIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico de Setúbal (Other)
Collaborators: Universidade Nova de Lisboa (Other)
Responsible Party: Principal Investigator, Eduardo B. Cruz, Principal Investigator Eduardo José Brazete Carvalho Cruz, Instituto Politécnico de Setúbal
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: SAICT-POL/23439
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Risk-stratification; STarT Back; Patient outcomes; Cost-effectiveness;; Barriers and Facilitators
MeSH Terms: conditions — Low Back Pain | interventions — Acetaminophen; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Other): All patients were referred for the study by their General Practitioner (GP). GPs were encouraged to assess and treat their patients as usual and make all the referrals they think are appropriate for their patients.
  Interventions: Drug: Usual Care
- Stratified Model of Care (Other): A subgrouping tool helps guide clinical decision-making about treatment and onward referral (Start Back Screening Tool). Patients in each subgroup (low, medium or high risk of chronicity) are then managed according to a targeted treatment system of increasing complexity.
  Interventions: Other: SPLIT Stratified Model of Care

INTERVENTIONS:
Drug: Usual Care — Pain Medication, imaging, referrals to other health services, other health care appointments
  Other Names: Pain Medication
  Arms: Usual Care
Other: SPLIT Stratified Model of Care — Physiotherapy targeted treatment system of increasing complexity for each subgroup (low, medium or high) of risk of chronicity. Includes patient education, manual therapy and exercise
  Other Names: Physiotherapy
  Arms: Stratified Model of Care

SUMMARY:
The SPLIT project evaluates the implementation of a stratified model of care for people with low back pain patients who consulted primary care.This involves evaluating the process of implementation as well as patient level outcomes.

The project consists of two phases: First, a before-after study comprising two sequential but independent cohort studies will be conducted to compare the outcomes and cost-effectiveness of current practice with the SPLIT stratified model of care. Second, an implementation strategy will be developed based on the results of a survey regarding determinants of current practice, and two focus groups concerning the barriers and facilitators for the implementation of the SPLIT stratified model of care.

DETAILED DESCRIPTION:
A before after study consisting of two sequential but independent cohorts of LBP patients, separated by a 3 months interval will be conducted in 6 primary care units in Portugal. In both cohorts participants will be recruited during a 7 months period.

Recruitment and data collection procedures will be identical for both cohorts. Participants will be eligible if they consult one of the participating General Practitioner practices (GA) due to non-specific Low Back Pain (LBP), with or without leg pain (The International Classification for Primary Care-2 diagnostic codes L03, L84, and L86), if they are aged between 18 and 65 years and able to read and speak the Portuguese language. They will be excluded if they have clinical signs of infection, tumor, osteoporosis, fracture, structural deformity, inflammatory disorder, radicular syndrome, or cauda equine syndrome, if they have severe depression or other psychiatric condition, if they are pregnant, or if they have undergone back surgery or conservative treatment in the prior 6 and 3 months, respectively.

Patients will be recruited by their GP, who will briefly explain the study and obtain consent to pass the contact details to a research assistant (RA). The RA will inform the patients about the study and ask them if they are willing to participate and to be contacted for follow-up questionnaires (by phone), and whether they give permission for their LBP medical records to be reviewed. Patients who decline referral will not be eligible for the study and will follow the usual clinical care.

On the initial screening with the RA, eligible LBP patients who consent to participate in the study will fill a questionnaire booklet containing socio-demographic and clinical questions, the Start Back Screening Tool, and patient reported outcomes concerning back-related disability (Roland Morris Disability Questionnaire), pain intensity (Numeric Pain Rating Scale), and health related quality of life (EuroQuol, five dimensions, 3 levels). These outcomes will be reassessed at 2 and 6 months following the first medical consultation. A Global Perceived Effect Scale (GPES) to assess patient overall perception of improvement with treatment will be added in the follow-up reassessments.

In both cohorts no specific instruction will be given to GPs concerning their practice. They will be encouraged to assess and treat their patients as usually and make all the referrals they think are appropriate for their patients. At the end of each cohort the GPs medical records will be reviewed and data concerning the number of primary care consultations, prescribed medications, ordering of diagnostic tests, referrals to other professionals or services will be extracted.

The primary outcome is back-related disability measured by the Roland Morris Disability Questionnaire (RMDQ). This questionnaire consists of 24 items related to activities of daily living and was developed to measure self-rated disability due to LBP. Each answer can be scored "0" or "1," thus leaving a range of scores from 0 to 24, with higher scores indicating higher disability. The RMDQ has shown good reliability, construct validity and responsiveness in studies with LBP patients. Secondary outcomes include pain, health related quality of life (HRQoL), and patients' perception of overall change of their back condition. Pain intensity will be measured by the Numeric Pain Rating Scale (NPRS). This is an 11-point self-report measure (0 to 10) with the labels "no pain" and "worst imaginable pain" on the ends, that has proven to be valid and reliable with patients with musculoskeletal pain. The EuroQuol, five dimensions, 3 levels (EQ-5D-3L) is a generic measuring instrument developed to assess HRQoL. The weight applied to the states is based on the Portuguese valuation study of the EQ-5D-3L. GPES is a transition scale designed to assess the patients' perception of overall change in their back condition. All patient reported measures are cross-culturally validated into European Portuguese Language showing adequate psychometric properties.

Two criteria will be used to interpret the response to treatment: 1) the Minimal Clinically Important Difference established for the RMDQ and NPRS (reduction of ≥30% from baseline); the definition of persisting LBP disability (RMDQ score >7) at 2 and 6 months.

In parallel with the data collection of the first cohort, an implementation plan will be developed. Determinants of practice (change) will be identified through the results of a survey about the GPs and Physical Therapists (PTs) attitudes, beliefs and confidence in managing LBP patients, and their adherence to clinical guidelines. Behavioural change strategies will be selected and implemented. Based on the published results of the current practice in primary care, and on the effectiveness of knowledge transfer strategies in similar studies, it is very likely that the intervention program will include different strategies such as patient-mediated interventions, educational meetings and key practice enablers (e.g. a web platform with information for patients, mentoring program, audit and feedback) targeted to GPs, PTs and patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Low back Pain of any duration;
* Age between 18 and 65 years;
* Able to read and speak the Portuguese language.

Exclusion Criteria:

* Clinical signs of infection;
* Clinical signs of tumor;
* Clinical signs of osteoporosis;
* Clinical signs of fracture;
* Clinical signs of structural deformity;
* Clinical signs of inflammatory disorder;
* Clinical signs of radicular syndrome;
* Clinical signs of cauda equine syndrome;
* Clinical signs of severe depression or other psychiatric condition;
* Pregnant women;
* Patients that undergone a back surgery in the prior 6 months;
* Patients that received any type of conservative treatment in the prior 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Low back Pain Disability will be assessed through the Roland Morris Disability Questionnaire (RMDQ) | Change on disability from baseline to 2 and 6 months
  The RMDQ consists of 24 items that measures the functional status over the past 24 hours in patients with LBP. Each answer can be scored "0" or "1", thus leaving a range of scores from 0 to 24, with higher scores indicating higher disability. The RMDQ has shown good validity and test-retest reliability with reported intraclass correlation coefficients (ICC) of 0.8 or more.

SECONDARY OUTCOMES:
Pain intensity will be assessed through the Numeric Pain Rating Scale (NPRS) | Change on pain intensity from baseline to 2 and 6 months
  Pain intensity will be measured with a numerical pain rating scale (NPRS). Participants were asked to rate the intensity of their current pain on a scale of 0 ("no pain") to 10 ("worst possible pain"). The NPRS has proven to be valid and reliable in patients with LBP pain. The NPRS will provide a score of pain intensity at the moment and in the last 4 weeks.
Health related Quality of life (HRQoL) will be assessed by the EuroQuol 5 dimensions, 3 levels (EQ-5D-3L) questionnaire. | Change on HRQoL from baseline to 2 and 6 months
  HRQoL will be measured with the Portuguese version of the EQ-5D-3L. The index of the health status of the individual, which varies from a higher value of "1" (corresponding to the best possible health), and "0" (death) will be calculated to assess HRQoL based on status in 5 dimensions: mobility, self-care, usual activities, pain discomfort and anxiety/depression, each with 3 levels of severity (0 = 'no problem', 1 = 'moderate problem', or 2 = 'extreme problem). The weight applied to the severity states will be based on the Portuguese valuation study of the EQ-5D-3L. Additionally the Health thermometer from EQ-5D-3L will be used (score 0= worst imaginable to 100= best imaginable) to assess the general health status.
Patients perception of global change will be assessed by the questionnaire Global Perceived Effect Scale | Global perception of change related with low back condition at 2 and 6 months follow-ups
  GPES is a transition scale designed to assess the patients' perception of change of their back condition. The GPES ranged from -5 ("vastly worse") to +5 ("completely recovered"). The GPES showed adequate test-rest reliability, validity and responsiveness. The GPES's score will be used to monitor the patient's global perception of change of his/ her low back condition.
Number of medical appointments for a low back pain complaint | The number of medical appointments concerning of each participant will be collected during the 6 months period after patient's enrollment
  The number of primary care visits to the General Practitioner for a low back pain complaint, for each participant, will be collected from local medical records.
The rate of imaging tests prescribed related with a low back pain complaint | The number of imaging tests prescribed will be collected during the 6 months period after patient's enrollment
  The number of x-rays, MRI and CT-scans of lower back will be collected for each participant from the local medical records.
The rate of pain medication for low back pain complaints | The low back pain medication will be collected during the 6 months period after patient's enrollment
  The name of the medication prescribed will be collected for each participant from the local medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Canhão, PhD, Study Chair — Epidoc Unit- Nova Medical School. Universidade Nova de Lisboa
Locations (1):
- Instituto Politécnico de Setúbal, Setúbal, Portugal

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will became available after publication which is anticipated for no earlier than 30 of June 2020. From this date, data will remain available for a period of 3 years.
Access Criteria: The data will be available on request.

REFERENCES:
- [Derived] Cruz EB, Canhao H, Fernandes R, Caeiro C, Branco JC, Rodrigues AM, Pimentel-Santos F, Gomes LA, Paiva S, Pinto I, Moniz R, Nunes C. Prognostic indicators for poor outcomes in low back pain patients consulted in primary care. PLoS One. 2020 Mar 27;15(3):e0229265. doi: 10.1371/journal.pone.0229265. eCollection 2020. PMID 32218561